CLINICAL TRIAL: NCT00634101
Title: The Comparative Clinical Performance of Narafilcon A and the FOCUS DAILIES AquaComfort Plus Lens
Brief Title: A Comparison of Two Daily Disposable Contact Lenses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was resurrected as NCT00727558 (CR-0808)
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0716; DISP-519
Record Dates: First submitted 2008-02-28; First posted 2008-03-12 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Refractive Error; Myopia
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- nefilcon A (Active Comparator): Subjects randomized to this arm received the nelfilcon A lens throughout the entire duration of the study.
  Interventions: Device: nelfilcon A
- narafilcon A (Experimental): Subjects randomized to this arm received the narafilcon A lens throughout the entire duration of the study.
  Interventions: Device: narafilcon A

INTERVENTIONS:
Device: nelfilcon A — contact lens
  Other Names: FOCUS DAILIES AquaComfort Plus
  Arms: nefilcon A
Device: narafilcon A — contact lens
  Other Names: Experimental Contact Lens
  Arms: narafilcon A

SUMMARY:
This study seeks to evaluate the clinical performance of a new CE marked daily disposable contact lens that contains a wetting agent to a recently improved daily disposable contact lens.

ELIGIBILITY:
Inclusion Criteria:

1. They are of legal age (18 years) and capacity to volunteer.
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They would be expected to attain at least 6/9 (20/30) in each eye with the study lenses.
5. They are able to wear contact lenses with a back vertex power of -1.00 to -6.00DS.
6. They have a maximum of 1.00D of refractive astigmatism (i.e. ≤ 1.00 DC).
7. They have successfully worn contact lenses within six months of starting the study.

Exclusion Criteria:

1. They have an ocular disorder which would normally contra-indicate contact lens wear.
2. They have a systemic disorder which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
7. They are pregnant or lactating.
8. They have grade 2 or greater of any of the following ocular surface signs: corneal oedema, corneal vascularisation, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
9. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV).
10. They have diabetes.
11. They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2008-03-01 (Actual); Study Completion 2008-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United Kingdom (20):
  - Simon Donne Opticians, Bedford, Bedfordshire
  - Brock & Houlford, Brislington, Bristol
  - Keith Tempany Opticians, Broadstone, Dorset
  - Cole Martin Tregaskis Optometrists, Brentwood, Essex
  - Specsavers Opticians, Colchester, Essex
  - Eyecare, Ilford, Essex
  - Cameron-Davies Optometrists, Southsea, Hants
  - Leightons Opticians, St Albans, Herts
  - Hazel Smith Opticians, Shanklin, Isle Of Wight
  - David Gould Opticians, Rawtenstall, Lancashire
  - Vision Express Optical Lab, Hendon, London
  - City Opticians, Holborn, London
  - David H. Burns, BSC, FCOptom, Tottenham, London
  - First Contact Opticians, Pinner, Middlesex
  - S.H. Harrold, Uxbridge, Middlesex
  - Dipple & Conway Opticians, Norwich, Norfolk
  - Tompkins Knight & Son, Northampton, Northamptonhsire
  - Chalmers & Sons (Opticians), Cardiff, South Glamorgan
  - Boots Opticians Ltd, Birmingham, West Midlands
  - Viewpoint, York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 129 subject were enrolled into this study. Of those enrolled, all were assigned to a study lens, however, only 125 eligble to be dispensed. Of those dispensed, 117 subjects completed the study. However, this study was utlimately terminated.
Groups:
- Test (Narafilcon A): Subjects randomized to receive the Test lens throughout the study
- Control (Nelfilcon A): Subjects randomized to receive the Control lens throughout the study
Period: Overall Study
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Started | 66 | 59
Completed | 61 | 56
Not Completed | 5 | 3
Not completed — Study Terminated | 3 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A) | Total
Number analyzed (Participants) | 67 | 62 | 129
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (10.4) | 33.9 (9.8) | 34.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 48 | 89
  Male | 26 | 14 | 40
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 67 | 62 | 129

OUTCOME MEASURES:

1. Primary Outcome: Comfort at the End of the Day
Description: Comfort at the end of the day was assessed by the individual questionnaire item "Comfort at the end of the day" with the response cateogries 1=Poor, 2=Fair, 3=Good, 4=Very good and 5=Excellent. EOD Comfort was also assessed by the individual item "How comfortable did your eyes feel at the end of the day when wearing the contact lenses you were provided?" with the respopnse categories of 1=Extremely Uncomfortable, 2=Very Uncomfortable, 3=Slightly Uncomfortable, 4=Comfortable and 5= Very Comfortable. The number of participants that responsed in each cateogry for each item was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Test (Narafilcon A): Subject that wore the Test lens throughout the study.
- Control (Nelfilcon A): Subject that wore the Control lens throughout the study.
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Comfort EOD: 5 | 8 | 7
  Comfort EOD: 4 | 17 | 12
  Comfort EOD: 3 | 10 | 15
  Comfort EOD: 2 | 5 | 8
  Comfort EOD: 1 | 13 | 7
  Comfort EOD: Intentionally Left Blank | 0 | 0
  Eye Comfort EOD: 5 | 14 | 7
  Eye Comfort EOD: 4 | 13 | 16
  Eye Comfort EOD: 3 | 14 | 18
  Eye Comfort EOD: 2 | 6 | 4
  Eye Comfort EOD: 1 | 6 | 3
  Eye Comfort EOD: Intentionally Left Blank | 0 | 1

2. Primary Outcome: Limbal Hyperaemia
Description: Limbal Hyperaemia was measured using Efron Grading Scale ranges from 0 to 4 with 0.5 units increments (0 = Normal, 1 = Trace, 2 = Mild, 3 = Moderate, 4 = Severe).
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 61 | 56
Number analyzed (eyes) | 122 | 112
eyes
  Grade 0 | 72 | 54
  Grade 0.5 | 26 | 34
  Grade 1 | 15 | 8
  Grade 1.5 | 0 | 8
  Grade 2 | 4 | 5
  Grade 2.5 | 4 | 3
  Grade 3 | 1 | 0
  Grade 3.5 | 0 | 0
  Grade 4 | 0 | 0

3. Secondary Outcome: Overall Handling
Description: Handling was assessed through opinion of handling in the final questionnaire. There were 5 categories Excellent (5), Very Good (4), Good (3), Fair (2) and Poor (1).
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 61 | 56
Participants
  Excellent (5) | 23 | 8
  Very Good (4) | 27 | 23
  Good (3) | 8 | 18
  Fair (2) | 3 | 6
  Poor (1) | 0 | 1

4. Primary Outcome: Comfort Immediately When You First Put Them on
Description: Comfort immediately when you first put them on was assessed by the individual questionnaire item "Comfort immediately when you first put them on" with the response cateogries 1=Poor, 2=Fair, 3=Good, 4=Very good and 5=Excellent. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Excellent (5) | 13 | 19
  Very Good (4) | 22 | 13
  Good (3) | 8 | 8
  Fair (2) | 6 | 7
  Poor (1) | 4 | 2

5. Primary Outcome: Comfort Throughout the Day
Description: Comfort throughout the day was assessed by the individual questionnaire item "Comfort throughout the day" with the response cateogries 1=Poor, 2=Fair, 3=Good, 4=Very good and 5=Excellent. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Excellent (5) | 13 | 19
  Very Good (4) | 22 | 13
  Good (3) | 8 | 8
  Fair (2) | 6 | 7
  Poor (1) | 4 | 2

6. Primary Outcome: Lack of Dryness at the End of the Day
Description: Lack of dryness at the end of the day was assessed by the individual questionnaire item "Not making your eyes feel dry even at the end of the day" with the response cateogries 1=Poor, 2=Fair, 3=Good, 4=Very good and 5=Excellent. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Excellent (5) | 12 | 9
  Very Good (4) | 11 | 12
  Good (3) | 9 | 8
  Fair (2) | 8 | 9
  Poor (1) | 13 | 9
  Intentionally left Blank | 0 | 2

7. Primary Outcome: Overall Opinion
Description: Overall opinion was assessed by the individual questionnaire item "Considering your experience with the contact lenses you were provided, which statement best describes your overall opinion of these contact lenses? " with the response cateogries 1=Poor, 2=Fair, 3=Good, 4=Very good and 5=Excellent. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Excellent (5) | 12 | 12
  Very Good (4) | 17 | 19
  Good (3) | 10 | 9
  Fair (2) | 9 | 8
  Poor (1) | 5 | 1

8. Primary Outcome: Overall Comfort
Description: Overall comfort was assessed by the individual questionnaire item "Overall Comfort" with the response cateogries 1=Poor, 2=Fair, 3=Good, 4=Very good and 5=Excellent. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Excellent (5) | 12 | 14
  Very Good (4) | 20 | 17
  Good (3) | 8 | 8
  Fair (2) | 6 | 7
  Poor (1) | 7 | 3

9. Primary Outcome: My Lenses Stayed Moist
Description: My Lenses Stayed Moist was assessed by the individual questionnaire item "They stayed moist and smooth, even after long hours at the computer" with the response cateogries 1=Disagree Strongly, 2=Disagree Somewhat, 3=Neither Agree Nor Disagree, 4=Very Somewhat and 5=Agree Strongly. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Agree Strongly (5) | 8 | 11
  Agree Somewhat (4) | 18 | 11
  Neither Agree Nor Disagree (3) | 8 | 10
  Disagree Somewhat (2) | 8 | 8
  Disagree Strongly (1) | 11 | 9

10. Primary Outcome: I Forgot i Was Wearing Lenses Was
Description: I forgot i was wearing lenses was assessed by the individual questionnaire item "They made me forget that I was wearing contact lenses" with the response cateogries 1=Disagree Strongly, 2=Disagree Somewhat, 3=Neither Agree Nor Disagree, 4=Very Somewhat and 5=Agree Strongly. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Agree Strongly (5) | 12 | 16
  Agree Somewhat (4) | 16 | 15
  Neither Agree Nor Disagree (3) | 6 | 4
  Disagree Somewhat (2) | 13 | 8
  Disagree Strongly (1) | 6 | 6

11. Primary Outcome: Mainted Natural Moisture
Description: Mainted natural moisture was assessed by the individual questionnaire item "They maintained my eyes' own natural moisture" with the response cateogries 1=Disagree Strongly, 2=Disagree Somewhat, 3=Neither Agree Nor Disagree, 4=Very Somewhat and 5=Agree Strongly. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Agree Strongly (5) | 14 | 10
  Agree Somewhat (4) | 17 | 16
  Neither Agree Nor Disagree (3) | 7 | 10
  Disagree Somewhat (2) | 10 | 6
  Disagree Strongly (1) | 5 | 7

12. Primary Outcome: Comfort While Wearing Lenses in Heat/Air Conditioned Environments
Description: Comfort while wearing lenses in heat/air conditioned environments was assessed by the individual questionnaire item "How often are you comfortable while sitting under or near an air conditioning vent or heating vent " with the response cateogries 0=Not Applicable, 1=Always, 2=Frequently, 3=Occasionally, 4=Rarely and 5=never. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Not Applicable (0) | 7 | 8
  Always (1) | 15 | 11
  Frequently (2) | 16 | 12
  Occasionally (3) | 10 | 10
  Rarely (4) | 4 | 6
  Never (5) | 1 | 2

13. Primary Outcome: Dryness at the End of the Day
Description: Dryness at the end of the day was assessed by the individual questionnaire item "How dry did your eyes feel at the end of the day when wearing the contact lenses you were provided" with the response cateogries 1=Extremely Dry, 2=Very Dry, 3=Moderately Dry, 4=Slightly Dry and 5=Not Dry at All. The number of participants that responsed in each cateogry was reported.
Time Frame: 1-Week Follow-up
Population: All available data at the 1-Week follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
Number analyzed (Participants) | 53 | 49
Participants
  Not Dry at all (5) | 22 | 11
  Slightly Dry (4) | 19 | 18
  Moderately Dry (3) | 2 | 11
  Very Dry (2) | 6 | 6
  Extremely Dry(1) | 4 | 2
  Intentionally Left Blank | 0 | 1

ADVERSE EVENTS:
Time Frame: Throughout the duration of this study. Approximately 1 week per subject.
Groups:
- Test (Narafilcon A): Subject that were dispensed the Test lens throughout the study.
- Control (Nelfilcon A): Subject that were dispensed the Control lens throughout the study.
Arm/Group | Test (Narafilcon A) | Control (Nelfilcon A)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/59
Other Adverse Events (participants affected / at risk) | 0/66 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days